CLINICAL TRIAL: NCT03497715
Title: A Randomised, Single Dose, 5 Way Crossover, Open-label Adaptive Design, Gamma Scintigraphy Study Comparing the Disintegration Profile of Oral Ibuprofen Lysine 2 x 342 mg, Ibuprofen Sodium 2 x 256 mg, Ibuprofen Liquid Capsules 2 x 200 mg and Two Reference Formulations of Ibuprofen Acid 2 x 200 mg in Healthy Volunteers
Brief Title: Gamma Scintigraphy Study to Investigate Tablet Disintegration in Healthy Volunteers.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: On completion of part 1 it was felt that there would be no benefit in completing part 2
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL1401
Record Dates: First submitted 2018-03-19; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1 (Experimental): Treatment order: Ibuprofen liquid capsules, Ibuprofen sodium, Ibuprofen (Nurofen), Ibuprofen lysine, Ibuprofen (Wockhardt)
  Interventions: Drug: Ibuprofen lysine; Drug: Ibuprofen Sodium; Drug: Ibuprofen; Drug: Ibuprofen (Nurofen); Drug: Ibuprofen (Wockhardt)
- Experimental 2 (Experimental): Treatment order: Ibuprofen lysine, Ibuprofen (Wockhardt), Ibuprofen sodium, Ibuprofen (Nurofen), Ibuprofen liquid capsules
  Interventions: Drug: Ibuprofen lysine; Drug: Ibuprofen Sodium; Drug: Ibuprofen; Drug: Ibuprofen (Nurofen); Drug: Ibuprofen (Wockhardt)
- Experimental 3 (Experimental): Treatment order: Ibuprofen liquid capsules, Ibuprofen (Nurofen)1, Ibuprofen sodium, Ibuprofen (Wockhardt), Ibuprofen lysine
  Interventions: Drug: Ibuprofen lysine; Drug: Ibuprofen Sodium; Drug: Ibuprofen; Drug: Ibuprofen (Nurofen); Drug: Ibuprofen (Wockhardt)
- Experimental 4 (Experimental): Treatment order: Ibuprofen (Wockhardt), Ibuprofen (Nurofen), Ibuprofen lysine, Ibuprofen liquid capsules, Ibuprofen sodium
  Interventions: Drug: Ibuprofen lysine; Drug: Ibuprofen Sodium; Drug: Ibuprofen; Drug: Ibuprofen (Nurofen); Drug: Ibuprofen (Wockhardt)

INTERVENTIONS:
Drug: Ibuprofen lysine — Test 1
  Other Names: Nurofen Migraine pain
Drug: Ibuprofen Sodium — Test 2
  Other Names: Nurofen Express
Drug: Ibuprofen — Test 3
  Other Names: Nurofen Immedia
Drug: Ibuprofen (Nurofen) — Reference 1
  Other Names: Nurofen
Drug: Ibuprofen (Wockhardt) — Reference 2

SUMMARY:
The study will be an adaptive, 2 part, single dose, 5-way crossover gamma scintigraphy study in healthy subjects, to investigate the rate and site of tablet disintegration of various forms of Ibuprofen.

DETAILED DESCRIPTION:
Ibuprofen is a non-steroidal anti-inflammatory drug (NSAID) with anti-inflammatory, analgesic and anti-pyretic properties. There are now a wide variety of formulations of ibuprofen available on market in which the active ingredient, ibuprofen, is either as the free acid, salt or salt in situ. As a result of differences between these formulations, differences in absorption and time to effectiveness are achieved. Rates of absorption are commonly assessed using pharmacokinetic (PK) studies, where the time taken for therapeutic plasma concentration levels to be reached can be determined, with associated absorption profiles being generated.

Before absorption can occur the product must disintegrate in the stomach and empty into the small intestine. Gamma scintigraphy may be used to assess the disintegration rate (of tablets/capsules/caplets) by acquiring images of the investigational medicinal product (IMP) in vivo. Through the use of radiolabelled dosage forms, it enables the visualisation of key stages preceding absorption, including tablet disintegration and the rate of gastric emptying. The assessment of these stages, which are required prior to absorption in the small intestine, may be useful in gaining an understanding of the differences between the dosage forms. The main purpose of this study is to visualise and determine the rate of disintegration and subsequent availability for absorption of different ibuprofen formulations, by gamma scintigraphy.

The study will be conducted in two parts. Part 1 will be conducted as a pilot phase where each subject will receive all 5 IMPs over 5 treatment visits (one IMP/visit).

The data generated in Part 1 will be assessed and used to determine whether to continue to Part 2 as planned, continue to Part 2 with adaptations or stop the study. Adaptations may involve altering the radiolabelling procedure and/or the gamma scintigraphy procedure and/or associated time-points and/or redefining primary/secondary endpoints and statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 18 to < 50 years.
2. Sex: Male.
3. Status: Healthy volunteers.

Exclusion Criteria:

1. A history of significant disease of any body-system.
2. Any condition that may currently interfere with the absorption, distribution, metabolism or excretion of drugs.
3. A history of allergy or intolerance (including angio-oedema, urticaria, bronchospasm and rhinitis) related to treatment with ibuprofen or other nonsteroidal anti-inflammatory drugs (NSAIDs) or the excipients of the formulations.
4. A history of peptic or duodenal ulcers or gastro-intestinal bleed or upper gastrointestinal bleed, or other significant gastro-intestinal disorders.
5. A history of frequent dyspepsia, e.g., heartburn or indigestion.
6. A history of migraine.
7. A history of psychotic illness, attempted suicide or parasuicide.
8. Current smokers and ex-smokers who have smoked within 6 months.
9. A history of drug abuse (including alcohol).
10. High consumption of stimulating drinks (coffee, tea, cola, energy drinks etc.; total caffeine intake per day above 300 mg (1 cup of coffee equates to 50 mg).
11. Those with positive drugs of abuse screen including alcohol on any occasion throughout the study.
12. Ingestion of a prescribed drug at any time in the 14 days before dosing with study medication (excluding hormonal contraceptives and hormone replacement therapy), or consumption of enzyme inhibitors or inducers during the previous month (such as barbiturates, carbamazepine, erythromycin, phenytoin, etc.).
13. Ingestion of an over-the-counter preparation within 7 days before dosing with study medication, including herbal medications, vitamin/fish oil supplements, ibuprofen and other NSAIDs and paracetamol.
14. Known human immune deficiency virus (HIV) positive status, or a positive viral serology screen.
15. Those unable in the opinion of the Investigator to comply fully with the study requirements.
16. Those who are unwilling to consume gelatin of animal origin.
17. Those previously randomised into this study.
18. Employee at study site.
19. Partner or first degree relative of the investigator
20. Those who have participated in a clinical trial in the previous 12 weeks.
21. Participation in a study in which radioisotopes were administered or in which subjects were exposed to any radiation (e.g. x-rays, handling of radiolabelled materials) other than normal background radiation within the 12 months before the screening visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 6 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Radioactive counts | 3 hours
  radioactivity counts as determined by gamma scintigraphy imaging